CLINICAL TRIAL: NCT03657329
Title: Performance of a Wireless Dry-EEG Device for Sleep Monitoring Compared to a Gold Standard Polysomnography in Patients With Suspected Sleep-Disordered Breathing
Brief Title: Comparison of Dreem to Clinical PSG for Sleep Monitoring in Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dreem (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTAVE Stanford
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Sleep; Sleep Apnea
Keywords: Automated Sleep Staging; Automated Apnea Detection
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Dreem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspicion of sleep-disordered breathing (Experimental): Dreem
  Interventions: Diagnostic Test: Dreem

INTERVENTIONS:
Diagnostic Test: Dreem — Dreem Band to be worn by each participant while undergoing in-lab sleep study with PSG. Pursuant to the physician-ordered diagnostic study, clinical staff may determine a split-night study with CPAP to be appropriate for any participant, simultaneous with the PSG and Dreem.

SUMMARY:
This study aims to evaluate the accuracy of apnea detection and automated sleep analysis by the Dreem dry-EEG headband and deep learning algorithm in comparison to the consensus of 5 sleep technologists' manual scoring of a gold-standard clinical polysomnogram (PSG) record in adults during a physician-referred overnight sleep study due to suspicion of sleep-disordered breathing.

DETAILED DESCRIPTION:
The study will enroll up to 70 adults who are referred to the Stanford Sleep Medicine Center by their physician for an overnight polysomnographic sleep study due to suspicion of sleep-disordered breathing, with the aim of collecting 60 usable data sets (i.e., eligible subjects with high-quality PSG and Dreem recordings). Upon arrival to the clinic, patients provide informed consent, are interviewed to determine eligibility, and complete a detailed demographic, medical, health, sleep, and lifestyle questionnaire (Alliance Sleep Questionnaire; ASQ). After the ASQ, participants are fitted with the PSG and the Dreem headband by the sleep technologist. During the PSG sleep study, the Dreem headband records EEG, pulse, oxygen saturation (SO2), movement, and respiratory rate. Many participants may undergo a split-night study with a continuous positive airway pressure (CPAP) device during their participation, as deemed necessary by the clinical staff pursuant to the sleep study.

The PSG data from the first 30 eligible participants will be manually scored by 5 sleep technologists. These manually-scored PSG data files (referred to as the training dataset) will be synchronized with Dreem data files from the same night and the synchronized files will be used to train Dreem's deep learning algorithms. Following training, the algorithms will be deployed to automatically score the final 30 participants' Dreem datasets (testing dataset). Finally, PSG records for the second 30 participants will be provided to the sponsor and manually scored by 5 sleep technologists. The manual scoring results will be compared to the Dreem automatic analysis to determine the accuracy of Dreem's apnea-hypopnea index (AHI) severity detection and sleep staging algorithms.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Capable of providing informed consent
* Suspicion of sleep breathing disorder (both diagnostic and split-night studies)

Exclusion Criteria:

* Concomitant diagnosis of a sleep disorder other than sleep apnea syndrome or insomnia
* Morbid obesity (BMI > 39)
* Use of benzodiazepines, nonbenzodiazepine (Z-drugs), or Gammahydroxybutyrate (GHB) the day/night of the study
* Concomitant diagnosis of cardiopulmonary or neurological comorbidities (such as heart failure, COPD, neurodegenerative conditions)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) severity agreement | Day 1
  AHI severity (normal [<5], mild [5-14], moderate [15-29], severe [>29]) as automatically determined by the Dreem headband compared to the AHI severity determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.

SECONDARY OUTCOMES:
Total Sleep Time (TST) agreement | Day 1
  Total time (in minutes) the subject spends asleep as automatically determined by the Dreem headband compared to the TST determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
EEG Virtual Channel signal quality agreement | Day 1
  Comparison of a proprietary signal quality metric between Dreem and PSG virtual channel, calculated as a ratio of supra-threshold quality signal time over total time in bed trying to sleep (lights off to lights on).
Wake After Sleep Onset (WASO) time agreement | Day 1
  Total time (in minutes) the subject spends awake from sleep onset to sleep end as automatically determined by the Dreem headband compared to the WASO determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N1 sleep stage agreement | Day 1
  Total time (in minutes) the subject spends in AASM N1 sleep stage as automatically determined by the Dreem headband compared to the N1 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N2 sleep stage agreement | Day 1
  Total time (in minutes) the subject spends in AASM N2 sleep stage as automatically determined by the Dreem headband compared to the N2 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N3 sleep stage agreement | Day 1
  Total time (in minutes) the subject spends in AASM N3 sleep stage as automatically determined by the Dreem headband compared to the N3 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in REM sleep stage agreement | Day 1
  Total time (in minutes) the subject spends in AASM REM sleep stage as automatically determined by the Dreem headband compared to the REM time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel H During, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Medicine Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share de-identified physiological data in an open-source format to the public. However, this will only occur if the data files are of sufficient quality and likely to be of use to the scientific community. This decision may also depend on certain legal or business constraints.